CLINICAL TRIAL: NCT05763329
Title: A Randomized, Double-blind, Placebo-Controlled Trial on the Effects of Lemborexant as a Treatment for Moderate-to-severe OSA Patients With Low Arousal Threshold
Brief Title: Effects of Lemborexant as a Treatment for Moderate-to-severe OSA Patients With Low Arousal Threshold
Acronym: LOSALAT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 218/64
Record Dates: First submitted 2023-02-09; First posted 2023-03-10 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-02

CONDITIONS: OSA
Keywords: Apnea/Hypopnea Index (AHI); Lemborexant; Obstructive Sleep Apnea (OSA); Low Arousal Threshold; Polysomnography
MeSH Terms: conditions — Apnea; Sleep Apnea, Obstructive | interventions — lemborexant; Tablets

STUDY DESIGN:
Intervention Model Description: The patients will be subsequently randomized 1:1 to one of the two treatment sequences. Participants will complete two overnight sleep studies and cross-over with 1-week wash-out period. Patients will receive either Lemborexant 5 mg per day or placebo prior 5 minutes before lights-out. Time of lights out was calculated from the median usual bedtime for each participant from the most recent 5 days (± 1 hour) and was kept constant between the two study nights. During this 2-night polysomnography, sleep parameters will be analyzed. The OSLER test to define vigilance will be obtained on the following morning.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lemborexant (Experimental): Patients will receive two treatment sequences. Participants will complete two overnight sleep studies and cross-over with 1-week wash-out period The participants will receive Lemborexant 5 mg per day 5 minutes before lights-out for one dose for the first overnight sleep test of the experiment. After 1 week wash-out period, the participants will cross to the placebo arm and receive placebo 5 minutes before lights-out for one dose for the second overnight sleep test of the experiment.
  Interventions: Drug: Lemborexant 5 MG Oral Tablet [Dayvigo] Day 1; Drug: Placebo Day 2
- Placebo (Placebo Comparator): Patients will receive two treatment sequences. Participants will complete two overnight sleep studies and cross-over with 1-week wash-out period The participants will receive placebo 5 minutes before lights-out for one dose for the first overnight sleep test of the experiment. After 1 week wash-out period, the participants will cross to the Lemborexant arm and receive Lemborexant 5 mg per day 5 minutes before lights-out for one dose for the second overnight sleep test of the experiment.
  Interventions: Drug: Lemborexant 5 MG Oral Tablet [Dayvigo] Day 2; Drug: Placebo Day 1

INTERVENTIONS:
Drug: Lemborexant 5 MG Oral Tablet [Dayvigo] Day 1 — Patients will receive Lemborexant 5 mg per day on the first day of sleep test
  Arms: Lemborexant
Drug: Lemborexant 5 MG Oral Tablet [Dayvigo] Day 2 — Patients will receive Lemborexant 5 mg per day on the second day of sleep test
  Arms: Placebo
Drug: Placebo Day 1 — Patients will receive placebo on the first day of sleep test
  Arms: Placebo
Drug: Placebo Day 2 — Patients will receive placebo on the second day of sleep test
  Arms: Lemborexant

SUMMARY:
The goal of this randomized, placebo-controlled, double-blind, crossover trial (1-week wash out period) is to compare 1 night of 5 mg Lemborexant to placebo administered before sleep in 10 moderate to severe OSA patients with low arousal threshold

The main questions it aims to answer are:

1. The effect of Lemborexant on apnea/hypopnea index (AHI) in moderate-to-severe OSA patients with low arousal threshold.
2. The effect of Lemborexant on the following parameters in moderate-to-severe OSA patients with low arousal threshold.

   * Arousal threshold
   * Mean and nadir oxygen saturation
   * Sleep latency
   * Sleep efficiency
   * Wake after sleep onset (WASO)
   * Percentage of time spent in NREM stage 1-3 and REM stage
   * Stanford Sleepiness Scale Questionnaire in the morning
   * The Oxford Sleep Resistance Test (OSLER) test

Participants will

* complete two overnight in-laboratory polysomnography (1-week washout)
* complete the OSLER test in the morning of the two overnight test

Researchers will compare with the placebo group to see if there is a difference in AHI

DETAILED DESCRIPTION:
Research Design A randomized, placebo-controlled, double-blind, crossover trial (1-week wash out period) comparing 1 night of 5 mg Lemborexant to placebo administered before sleep.

Research Methodology Participants A total of 10 moderate to severe OSA patients with low arousal threshold are randomized 1:1 to either Lemborexant or placebo. The participants will complete two overnight in-laboratory polysomnography (1-week washout). Next-morning alertness will also be assessed using OSLER test, respectively.

Inclusion criteria

Eligible, healthy individuals with all the followings:

* Untreated OSA patient 18 - 65 years of age
* AHI ≥15 events/h of sleep
* Low arousal threshold

Study protocol All patients who were previously diagnosed with moderate to severe obstructive sleep apnea from baseline polysomnography with a low arousal threshold will be enrolled.

The patients will be subsequently randomized 1:1 to one of the two treatment sequences. Participants will complete two overnight sleep studies and cross-over with 1-week wash-out period. Patients will receive either Lemborexant 5 mg per day or placebo prior 5 minutes before lights-out.

During this 2-night polysomnography, sleep parameters will be analyzed including AHI, mean and nadir oxygen indices, sleep latency, sleep efficiency, wake after sleep onset (WASO), and percentage of time spent in NREM, stage 1-3 and REM stage. The OSLER test to define vigilance will be obtained on the following morning.

ELIGIBILITY:
Inclusion Criteria:

* Untreated OSA patient 18 - 65 years of age(49)
* AHI ≥15 events/h of sleep (moderate to severe)(23, 49)
* Low arousal threshold was defined using previously recommended criteria which allocated a score of 1 to each criterion that was satisfied: (apnea-hypopnea index, <30 events per hour) + (nadir oxygen saturation as measured by pulse oximetry >82.5%) + (fraction of hypopneas >58.3%). A score of 2 or above defined a low arousal threshold(50) (low arousal threshold defined as esophageal pressure values are 0 to -15 cmH2O)(27)

Exclusion Criteria:

* Previous allergy or adverse effects with Lemborexant or other sedatives - Taking any medication that affects sleep or other variable measured in this study - Pregnant or nursing mothers - Respiratory disorders other than OSA - Comorbid disease of poor controlled or resistant hypertension, uncontrolled cardiovascular or cerebrovascular disease
* Using CPAP or other dental devices
* Unable to tolerate equipment in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
apnea/hypopnea index (AHI) | through study completion, one week
  AHI

SECONDARY OUTCOMES:
Mean and nadir oxygen saturation | through study completion, one week
Sleep latency (Time the patients fall asleep) | through study completion, one week
  Time spent from light out to the first 20 consecutive 30-second period of nonwakefulness (minutes)
Sleep efficiency (Time the patients actually sleep through out the experiment) | through study completion, one week
  Time the patient sleep per time in bed which is the total sleep time per time from light out until light on (total record time (TRT) (8 hours) (minutes)
Wake after sleep onset (WASO) | through study completion, one week
  Total time of wakefulness after initial sleep onset until light on
Percentage of time spent in NREM stage 1-3 and REM stage | through study completion, one week
The Oxford Sleep Resistance Test (OSLER) test | through study completion, one week

CONTACTS AND LOCATIONS:
Overall Officials: Sarocha Vivatvakin, MD, Principal Investigator — Department of Medicine, Faculty of Medicine, Chulalongkorn University
Locations (1):
- Chulalongkorn University, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No